CLINICAL TRIAL: NCT01029405
Title: A Double-Blind,Randomized, 12 Week, Bilateral Study of the Safety and Efficacy of AN2728 Ointment B, 2% and 0.5%, Versus Ointment B Vehicle in the Treatment of Patients With Plaque Type Psoriasis
Brief Title: Safety and Efficacy Study of a Novel Ointment to Treat Plaque Type Psoriasis
Acronym: AN2728PSR203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2728-PSR-203; C3291016 (Other: Pfizer)
Record Dates: First submitted 2009-12-07; First posted 2009-12-10 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Psoriasis
Keywords: Topical; Plaque type psoriasis
MeSH Terms: conditions — Psoriasis | interventions — crisaborole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1. AN2728 Ointment B (Active Comparator): 2%, administered twice daily
  Interventions: Drug: AN2728
- 2. AN2728 Ointment B Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo
- 3. AN2728 Ointment B (Active Comparator): 2%, administered once daily
  Interventions: Drug: AN2728
- 4. AN2728 Ointment B (Active Comparator): 0.5%, administered twice daily
  Interventions: Drug: AN2728
- 5. AN2728 Ointment B (Active Comparator): 0.5%, administered once daily
  Interventions: Drug: AN2728

INTERVENTIONS:
Drug: AN2728 — Ointment B, 2% or 0.5% applied once or twice daily
  Arms: 1. AN2728 Ointment B; 3. AN2728 Ointment B; 4. AN2728 Ointment B; 5. AN2728 Ointment B
Drug: Placebo — Ointment B Vehicle applied once or twice daily
  Arms: 2. AN2728 Ointment B Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AN2728 Ointment B, 2.0% and 0.5%, compared to Ointment Vehicle B, applied once or twice daily for 12 weeks, in the treatment of plaque type psoriasis

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, vehicle-controlled, bilateral design. Patients will apply both test article AN2728 Ointment B (0.5% or 2%), and Ointment B Vehicle twice daily for 12 weeks. The assigned study medication will be applied to two comparable treatment targeted plaques identified at baseline. One test article will be applied to one plaque and the other test article to an anatomically distinct plaque. All efficacy evaluations will be measured from only the two plaques identified at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age at time of enrollment
* Clinical diagnosis of stable plaque type psoriasis
* Two target plaques of similar severity meeting the following criteria:

  * 5 cm2 and ≤ 100 cm2, computed by multiplying the greatest diameter of the plaque by the diameter of the plaque perpendicular to the greatest diameter Bilaterally located (right/left) plaques on the arms or plaques located on the trunk. Plaques located on the trunk must be separated by at least 10 cm Overall target plaque severity score (OTPSS) of 2-4 (mild to moderate) with no more than a 1 point difference in the scores of the two target plaques
* Willing and able to apply study drug as directed, comply with study instructions and commit to all follow-up visits
* Ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol related procedures

Exclusion Criteria:

* Any dermatological conditions, disease state or physical condition that could interfere with clinical evaluations or might expose the patient to an unacceptable risk by study participation
* Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy (see below)
* Clinically significant, abnormal Screening laboratory results (unless approved by the medical monitor)
* Known sensitivity to any of the components of the study medication
* Spontaneously improving or rapidly deteriorating psoriatic plaques or pustular/exfoliative, guttate, erythrodermic or other non-plaque form of psoriasis
* Concomitant use of topical or systemic therapies that might alter the course of psoriasis
* Females of child bearing potential. Females must be post-menopausal (based on FSH levels) or surgically sterile (hysterectomy or bilateral oophorectomy)
* Washout periods for exclusionary therapies:

Oral retinoids: 8 weeks Non-retinoid systemic drugs that might alter the course of psoriasis: 4 weeks Psoralens with UV-A (PUVA): 4 weeks Ultraviolet-B (UVB) therapy: 4 weeks Topical drugs that might alter the course of psoriasis: 2 weeks Use of emollients/moisturizers on area(s) to be treated: 2 days prior to Baseline visit

* AIDS or AIDS-related illness
* Concurrent participation in another drug or device research study or within 30 days prior to enrollment
* Use of lithium- or hydroxychloroquine-containing products (e.g., Plaquenil)
* Use of a beta-blocking medication (e.g., Propranolol) if the dose has not been stabilized for at least 3 months
* Use of AN2728 in a previous clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Mexico (5):
  - Chihuahua City, Chihuahua
  - Mexico City, D.f.
  - Zapopan, Jalisco
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potosí

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2728 Ointment B 0.5 Percent + Ointment B Vehicle, Once Daily: AN2728 ointment B 0.5 percent (%) and ointment B vehicle was applied to 2 comparable and anatomically distinct treatment-targeted plaques respectively within each participant, once daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment B 0.5 Percent +Ointment B Vehicle, Twice Daily: AN2728 ointment B 0.5 percent and ointment B vehicle was applied to 2 comparable and anatomically distinct treatment-targeted plaques respectively within each participant, twice daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment B 2 Percent + Ointment B Vehicle, Once Daily: AN2728 ointment B 2 percent and ointment B vehicle was applied to 2 comparable and anatomically distinct treatment-targeted plaques respectively within each participant, once daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment B 2 Percent + Ointment B Vehicle, Twice Daily: AN2728 ointment B 2 percent and ointment B vehicle was applied to 2 comparable and anatomically distinct treatment-targeted plaques respectively within each participant, twice daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | AN2728 Ointment B 0.5 Percent + Ointment B Vehicle, Once Daily | AN2728 Ointment B 0.5 Percent +Ointment B Vehicle, Twice Daily | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Once Daily | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Twice Daily
Started | 36 | 37 | 35 | 37
Completed | 34 | 34 | 31 | 32
Not Completed | 2 | 3 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1 | 2
Not completed — Other | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all randomized participants who received the study medication.
Groups:
- AN2728 Ointment B 0.5 Percent + Ointment B Vehicle, Once Daily: AN2728 ointment B 0.5 percent and ointment B vehicle was applied to 2 comparable and anatomically distinct treatment-targeted plaques respectively within each participant, once daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
- Total: Total of all reporting groups
Arm/Group | AN2728 Ointment B 0.5 Percent + Ointment B Vehicle, Once Daily | AN2728 Ointment B 0.5 Percent +Ointment B Vehicle, Twice Daily | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Once Daily | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Twice Daily | Total
Number analyzed (Participants) | 36 | 37 | 35 | 37 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 1
  Between 18 and 65 years | 36 | 31 | 34 | 33 | 134
  >=65 years | 0 | 5 | 1 | 4 | 10
Gender [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 4 | 18
  Male | 30 | 33 | 31 | 33 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Greater Decrease In Overall Target Plaque Severity Score (OTPSS): Ointment (2% Twice Daily), Vehicle
Description: OTPSS is a scale to assess plaque severity. Each target plaque was scored by the investigator on severity scale ranging from 0 (no plaque) to 8 (very severe plaque), where higher score indicates more severity of a plaque. In this outcome measure, percentage of participants with reduced OTPSS in ointment (2% twice daily) treated plaque versus (vs.) vehicle treated plaque and percentage of participants with reduced OTPSS in vehicle treated plaque versus ointment (2% twice daily) treated plaque respectively at Day 42 are reported.
Time Frame: Day 42
Population: Intent-to-treat population included all randomized participants who received study medication.
Measure: Number; unit: percenatge of participants
Arm/Group | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Twice Daily
Number analyzed (Participants) | 37
percenatge of participants
  Ointment Treated Plaque vs. Vehicle Treated Plaque | 54.1
  Vehicle Treated Plaque vs. Ointment Treated Plaque | 2.7
Statistical Analysis 1: Comparison: AN2728 Ointment B 2 Percent + Ointment B Vehicle, Twice Daily; Test type: Superiority or Other; p < 0.001, 2-sided sign test

2. Secondary Outcome: Percentage of Participants With Greater Decrease In OTPSS: Ointment (0.5 % Once Daily, 0.5% Twice Daily and 2% Once Daily), Vehicle
Description: OTPSS is a scale to assess plaque severity. Each target plaque was scored by the investigator on severity scale ranging from 0 (no plaque) to 8 (very severe plaque), where higher scores indicated more severity of a plaque. In this outcome measure, percentage of participants with reduced OTPSS in ointment (0.5 % once daily, 0.5% twice daily and 2% once daily) treated plaque versus vehicle treated plaque and percentage of participants with reduced OTPSS in vehicle treated plaque versus ointment (0.5 % once daily, 0.5% twice daily and 2% once daily) treated plaque respectively at Day 42 are reported.
Time Frame: Day 42
Population: Intent-to-treat population included all randomized participants who received the study medication.
Measure: Number; unit: percenatge of participants
Arm/Group | AN2728 Ointment B 0.5 Percent + Ointment B Vehicle, Once Daily | AN2728 Ointment B 0.5 Percent +Ointment B Vehicle, Twice Daily | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Once Daily
Number analyzed (Participants) | 36 | 37 | 35
percenatge of participants
  Ointment Treated Plaque vs. Vehicle Treated Plaque | 30.6 | 43.2 | 40.0
  Vehicle Treated Plaque vs. Ointment Treated Plaque | 11.1 | 8.1 | 0.0

ADVERSE EVENTS:
Description: Adverse events were assessed in safety population which included participants who received study medication and provided a safety evaluation.
Arm/Group | AN2728 Ointment B 0.5 Percent + Ointment B Vehicle, Once Daily | AN2728 Ointment B 0.5 Percent +Ointment B Vehicle, Twice Daily | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Once Daily | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37 | 0/34 | 0/37
Other Adverse Events (participants affected / at risk) | 9/36 | 14/37 | 12/34 | 16/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AN2728 Ointment B 0.5 Percent + Ointment B Vehicle, Once Daily (N=36) | AN2728 Ointment B 0.5 Percent +Ointment B Vehicle, Twice Daily (N=37) | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Once Daily (N=34) | AN2728 Ointment B 2 Percent + Ointment B Vehicle, Twice Daily (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Swelling (General disorders) | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 3 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 0/30 | 0/33 | 1/30 | 0/33 — This adverse event was gender specific.
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.